CLINICAL TRIAL: NCT03561025
Title: Diagnostic Potential of PET/MRI in Cardiac Sarcoidosis: A Pilot Study Combining Advanced MRI and 18F-FDG and 18F-GE180 PET of the Myocardium
Brief Title: Diagnostic Potential of PET/MRI in Cardiac Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2016/883; 2017-000331-14 (EudraCT Number)
Record Dates: First submitted 2018-06-06; First posted 2018-06-19 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Sarcoidosis; Cardiomyopathies
Keywords: Diagnostic Imaging; Positron Emission Tomography Computed Tomography; Magnetic Resonance Imaging
MeSH Terms: conditions — Sarcoidosis; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18F-FDG-PET/MRI (Active Comparator)
  Interventions: Diagnostic Test: 18F-FDG-PET/MRI; Diagnostic Test: 18F-GE180-PET/MRI
- 18F-GE180-PET/MRI (Experimental)
  Interventions: Diagnostic Test: 18F-FDG-PET/MRI; Diagnostic Test: 18F-GE180-PET/MRI

INTERVENTIONS:
Diagnostic Test: 18F-FDG-PET/MRI — Contrast-enhanced MRI scanning after injection of 18F-FDG
Diagnostic Test: 18F-GE180-PET/MRI — Contrast-enhanced MRI scanning after injection of 18F-GE180

SUMMARY:
The aim of the study is to find better and more specific non-invasive methods to diagnose and stage cardiac sarcoidosis with the use of advanced imaging modalities, simultaneous 3T MRI and PET. Cardiac sarcoidosis is a disease of possibly fatal outcome in young people. The use of a combined PET/MRI system with 18F-FDG and a new inflammation-tracer (18F-GE180) can become a future game changer.

Sarcoid induced focal inflammation in myocardium should show high 18F-GE180 uptake. 18F-GE180 PET scans will give reliable data about inflammatory sarcoidosis activity in the myocardium. 18F-GE180 PET is expected to improve diagnostic accuracy compared to 18F-FDG-PET and/or contrast enhanced MRI.

ELIGIBILITY:
Inclusion Criteria:

* Heart department: Suspicion of myocardial sarcoidosis after contrast enhanced cardiac MRI
* Lung department: Clinically verified lung and/or mediastinal sarcoidosis

Exclusion Criteria:

* Known malignancies
* Treatment for sarcoidosis started
* Severe arrhythmia
* Patients with pacemakers or defibrillator
* Claustrophobia
* Known alcohol or drug abuse
* Kidney failure (eGFR < 30)
* Weight > 120 kg
* Diabetes Mellitus type I and II
* Patients that take immunosuppressive or immunomodulatory medication for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of a combined 18F-FDG and 18F-GE-180 PET/MRI examination for diagnosing cardiac sarcoidosis | One day after the test

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Søvik, Study Chair — St. Olavs Hospital
Locations (1):
- St Olav University Hospital, Dept Radiology and Nuclear Medicine, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided